CLINICAL TRIAL: NCT06744907
Title: Subdermal Betadine to Reduce Microbacterial Bioburden During Posterior Spinal Fusion
Brief Title: Safety and Efficacy of Subdermal Betadine During Posterior Spinal Fusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Lorena Floccari, Orthopedic Surgeon, Director Spine Center of Excellence, Director Spine Research, Akron Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-114
Record Dates: First submitted 2024-11-21; First posted 2024-12-20 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Spinal Fusion
Keywords: Spinal Fusion; Lumbar Spine; Thoracic Spine; Subdermal Betadine; Microbacterial bioburden

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10% Povidone-Iodine Arm (Active Comparator): A single-use sealed packet of three 10% povidone-iodine swabs will be opened via standard sterile technique. Three topical applications of 10% povidone-iodine along the length of the subdermis, using each of the 3 swab sticks provided from the sterile single-use packet. The solution will be allowed to dry at least three minutes. A culture will be obtained by rubbing an Eswab along the incision in the subdermis. Surgical exposure will proceed. After exposure is complete, an additional culture will be obtained with an Eswab in the deep wound. After corrective maneuvers are complete a final culture will be obtained with an Eswab just prior to wound closure.
  Interventions: Biological: 10% Povidone-Iodine Arm
- Saline Arm (Active Comparator): Three sterile swabs will be provided for soaking in sterile saline. Three applications of sterile saline along the length of the subdermis, using each of the 3 swabs soaked in sterile saline. The solution will be allowed to dry at least three minutes. A culture will be obtained by rubbing and Eswab along the incision in the subdermis. Surgical exposure will proceed. After exposure is complete, and additional culture will be obtained with and Eswab in the deep wound. After corrective maneuvers are complete a final culture will be obtained with and Eswab just prior to wound closure.
  Interventions: Procedure: Saline Arm

INTERVENTIONS:
Biological: 10% Povidone-Iodine Arm — A second application of surgical antisepsis with a topical povidone-iodine in the subdermal layer after making an incision.
  Arms: 10% Povidone-Iodine Arm
Procedure: Saline Arm — An application of saline in the subdermal layer after making an incision.
  Arms: Saline Arm

SUMMARY:
Bacterial in the subdermal layer of the skin, such as in hair follicles and sweat glands, may contaminate surgical wounds. The goal of this study is to learn about povidone-iodine and its ability to prevent infections specifically in patients with scoliosis receiving a spinal fusion.

DETAILED DESCRIPTION:
This is a prospective, one site, randomized controlled trial. The goal of this project is to evaluate the efficacy of subdermal 10% povidone-iodine at reducing bacterial contamination from the subdermal layer of skin during posterior spinal fusion. The primary outcome of this study will be incidence of positive bacterial growth in several layers of the surgical wound. Secondary outcomes will be complications, including allergic reactions, contact dermatitis, surgical site infection and wound complications. Finally, patient and surgical variables that can effect microbial growth will be observed.

Once identified, the surgeon and coordinators will discuss risks, benefits, advantages, and disadvantages of this study to eligible patients. If the family wishes to enroll, the patient's family and patient will be consented. And automatically randomized to either povidone-iodine vs control group (predetermined according to the statistician). All patients will follow the standardized spine pathway including standard antibiotics and skin preparation with isopropyl alcohol followed by ChloraPrepTM and sterile draping. Five bacterial cultures will be obtained throughout the spinal fusion similarly for all patients by rubbing along the entirety of the posterior spinal incision. The first two cultures will be taken before the placement of an antimicrobial adhesive drape and after the initial incision in the subdermal layer. The surgeon will be notified which group the patients are in. Patients who were randomized to the povidone-iodine group will then have three topical applications of 10% povidone-iodine along the length of the subdermis, using each of the 3 swab sticks provided from the sterile single-use packet. Patients who were randomized to the control group will then have three applications of sterile saline along the length of the subdermis, using each of the 3 swab sticks soaked in sterile saline. Following the 10% povidone-iodine or saline application, the solution will be allowed to dry at least three minutes and a third culture will be obtained. Surgical exposure will proceed in all patients, and an additional culture will be obtained along the length of the deep wound after exposure, and a final culture along the length of the deep wound just prior to wound closure. The swabs will be cultured, and the final results will be reported however, the surgeons delivering patient care will be blinded to the results to mitigate competing interests. Routine postoperative care will follow standard of care no matter the culture results. A data safety monitor will assure no correlation between culture results and infection rate.

ELIGIBILITY:
Inclusion Criteria

* Males and females
* Undergoing primary posterior spinal fusion of the thoracic and/or lumbar spine
* English Speaking

Exclusion Criteria

* Patients who have undergone prior spinal surgery
* Undergoing procedures other than primary posterior spinal fusion of the thoracic and/or lumbar spine (cervical fusion, anterior surgery, growth-friendly instrumentation)
* Any contraindication to povidone-iodine, including pregnancy, allergy, or prior treatment with radioiodine

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of bacterial growth in five layers of the surgical wound between the treatment group (10% povidone-iodine) and the control group (saline). | From enrollment to one year post operative.
  1. The skin, along the length of the planned incision
  2. The subdermis before application of povidone-iodine versus control with saline
  3. The subdermis after application of povidone-iodine versus control with saline)
  4. The deep surgical wound after exposure
  5. The deep surgical wound after all corrective maneuvers are complete, before closure

SECONDARY OUTCOMES:
To report the incidence of treatment-related and other adverse events, including allergic. | From enrollment to one year post operative.
  Secondary outcomes will be complications, including allergic reactions, contact dermatitis, surgical site infection and wound complications.

OTHER OUTCOMES:
To perform statistical correlations among locations/conditions and between treatment groups will be conducted in a generalized linear mixed model (GLMM) framework with a binomial distribution and a logit link function. | From enrollment to one year post operative.
  * Age
  * Gender
  * Comorbidities
  * Body mass index (BMI)
  * Operative time
  * Blood loss
  * Fusion levels
  * Scoliosis etiology
  * Curve type
  * Curve magnitude (Cobb angle)
  * Use of prophylactic antibiotics
  * Hospital length of stay
  * Complications, including readmissions and reoperations.

CONTACTS AND LOCATIONS:
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT06744907/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT06744907/ICF_001.pdf